CLINICAL TRIAL: NCT03085680
Title: Does Dietary Supplementation With Curcumin Maintain or Improve Physical and Cognitive Function in Aging Adults at Increased Risk for Disability?
Brief Title: Curcumin and Function in Older Adults
Acronym: SPICE
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: National Institute on Aging (NIA) (NIH); National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: IRB201600334-N; P30AG028740 (NIH); IRB201701371 (Other: UF Ancillary Study ID)
Record Dates: First submitted 2017-03-15; First posted 2017-03-21 (Actual); Results first posted 2022-02-02 (Actual); Last update posted 2022-07-26 (Actual); Status verified 2022-07

CONDITIONS: Older Adults; Physical Function; Cognitive Function
Keywords: Curcumin, physical function, cognitive function
MeSH Terms: interventions — Curcumin; microcrystalline cellulose

STUDY DESIGN:
Intervention Model Description: Randomized placebo-controlled design.
Who Masked: Participant, Investigator
Masking Description: Double-blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Curcumin (Experimental): Participants will be given identical capsules containing curcumin (1000 mg/day), and will be instructed to consume two 500 mg capsules prior to breakfast every morning with a glass of water. Participants will be instructed to follow this dosing regimen throughout the entire three-month treatment period. Compliance with the dosing regimen will be monitored both through interview and by counting capsules left at monthly clinic visits.
  Interventions: Drug: Curcumin
- Placebo (Placebo Comparator): Participants will be given identical capsules containing placebo (microcrystalline cellulose) and will be instructed to consume two 500 mg capsules prior to breakfast every morning with a glass of water. Participants will be instructed to follow this dosing regimen throughout the entire three-month treatment period. Compliance with the dosing regimen will be monitored both through interview and by counting capsules left at monthly clinic visits.
  Interventions: Drug: microcrystalline cellulose

INTERVENTIONS:
Drug: Curcumin — Participants will be given curcumin (1000 mg/day), and will be instructed to consume two 500 mg capsules prior to breakfast every morning with a glass of water. Participants will be instructed to follow this dosing regimen throughout the entire three-month treatment period. Compliance with the dosing regimen will be monitored both through interview and by counting capsules left at monthly clinic visits.
  Other Names: Turmeric; C3 Complex
  Arms: Curcumin
Drug: microcrystalline cellulose — Participants will be instructed to consume two capsules prior to breakfast every morning with a glass of water. Participants will be instructed to follow this dosing regimen throughout the entire three-month treatment period. Compliance with the dosing regimen will be monitored both through interview and by counting capsules left at monthly clinic visits.
  Other Names: placebo
  Arms: Placebo

SUMMARY:
This placebo-controlled RCT tests whether dietary supplementation with curcumin maintains or improves cognitive and physical function in older adults who are at high risk of functional decline due existing (mild) functional impairments and elevated biomarkers of inflammation and explore the association between functional changes and changes in biological indicators of active inflammation.

ELIGIBILITY:
Inclusion Criteria:

* Age > 65 years
* Usual walking speed <1 m/sec and >0.44 m/sec on the 4 m walk
* Sedentary lifestyle (< 120 min per week of moderate intensity physical activity);
* CRP > 1.0 mg/dL
* Willingness and ability to give informed consent
* Willingness to be randomized to the intervention groups
* Availability for participation through duration of study

Exclusion Criteria:

Exclusion Criteria (General)

* Unable to complete 400 meter walk test
* Failure or inability to provide informed consent
* Residence in a Skilled Nursing Facility (SNF); residence in an Assisted Living Facility (ALF) or independent housing is allowed
* Self-reported inability to walk one block
* Blood pressure readings >160/100
* Significant cognitive impairment, defined as a known diagnosis of dementia, or a Mini-Mental State Exam (MMSE) score <24
* Unable to communicate because of severe hearing loss or speech disorder
* Clinically significant depression (CES-D score > 20)
* Severe cardiac disease, including NYHA Class III or IV congestive heart failure, clinically significant aortic stenosis, history of cardiac arrest, use of a cardiac defibrillator, or uncontrolled angina
* Severe pulmonary disease, pneumonitis or interstitial lung disease
* Severe rheumatologic or orthopedic diseases (e.g., awaiting joint replacement, active inflammatory disease)
* Neurological conditions that cause impaired muscle function or mobility (e.g., Parkinson's Disease, multiple sclerosis, ALS)
* Other significant co-morbid medical disease (e.g. renal failure with eGFR < 30 ml/minute or on hemodialysis) or severe psychiatric disorder (e.g. bipolar, schizophrenia)
* Terminal illness with life expectancy less than 12 months, as determined by a physician
* Excessive alcohol use, defined as more than 5 drinks/day for males or more than 4 drinks/day for females, or more than 14 drinks per week
* Current smoker or less than 3 years smoking cessation
* Participating in another clinical trial or receiving an investigational product within 3 months prior to screening/enrollment

Exclusion Criteria (Curcumin-related)

* Diabetes mellitus currently taking medications to lower blood glucose (oral or by injection)
* Current use of anticoagulant or anti-platelet medications (aspirin 81 mg daily is allowed)
* Congenital or acquired bleeding disorders
* Cholelithiasis or other gall bladder or biliary tract disease
* Chronic gastrointestinal blood loss or iron deficiency (serum ferritin < 12 ng/mL, with or without anemia)
* History of estrogen-sensitive conditions including breast, uterine, and ovarian cancers; endometriosis; and uterine fibroids
* History of Tuberculosis (TB), HIV, Hepatitis B or C, or other disease potentially compromising immune function
* Current use of medications targeting immune or inflammatory function (e.g., sulfasalazine)
* Current use of anabolic medications (i.e., growth hormones or testosterone), antidepressant medications and antipsychotic agents (including monoamine oxidase inhibitors), or anticholinesterase inhibitors (i.e., Aricept)

Temporary Exclusion Criteria

* Acute infection (urinary, respiratory, other) or hospitalization within 1 month
* Myocardial infarction, CABG, or valve replacement within past 6 months
* Pulmonary embolism or deep venous thrombosis within past 6 months
* Stroke, hip fracture, hip or knee replacement, or spinal surgery within past 4 months
* Receiving physical therapy for gait, balance, or other lower extremity training

Ages: 65 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 17 (Actual)
Dates: Start 2017-08-11 (Actual); Primary Completion 2019-10-18 (Actual); Study Completion 2019-10-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephen D Anton, PhD, Principal Investigator — University of Florida
Locations (1):
- University of Florida, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Curcumin | Placebo
Started | 9 | 8
Completed | 9 | 8
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Curcumin | Placebo | Total
Number analyzed (Participants) | 9 | 8 | 17
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 9 | 8 | 17
Age, Continuous [Mean (Standard Deviation); unit: Years] | 79.4 (10.1) | 76.2 (5.6) | 77.8 (7.85)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 4 | 8
  Male | 5 | 4 | 9
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 9 | 8 | 17
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 9 | 8 | 17

OUTCOME MEASURES:

1. Primary Outcome: Curcumin and Physical Function -Walking
Description: To examine the effects of dietary supplementation with curcumin on changes in physical function walking speed- 400meter walk test.
Time Frame: Change in walking speed (meters/second) from Baseline and 3 months
Measure: Mean (Standard Deviation); unit: meters/second
Arm/Group | Curcumin | Placebo
Number analyzed (Participants) | 9 | 8
meters/second | 0.014 (0.090) | 0.103 (0.10)

2. Primary Outcome: Curcumin and Physical Function - Hand Grip
Description: To examine the effects of dietary supplementation with curcumin on changes in physical function grip strength- hand dynamometer
Time Frame: Change in grip strength (kilograms) from Baseline and 3 months
Measure: Mean (Standard Deviation); unit: Kilograms
Arm/Group | Curcumin | Placebo
Number analyzed (Participants) | 9 | 8
Kilograms | 0.63 (4.90) | -0.25 (3.14)

3. Secondary Outcome: Curcumin and Cognitive Function - Attention & Memory
Description: To examine the effects of dietary supplementation with curcumin on cognitive performance mini-mental state examination. 30 points max. The lower, the worse score.
Time Frame: Change in attention from Baseline and 3 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Curcumin | Placebo
Number analyzed (Participants) | 9 | 8
units on a scale | 0.33 (3.94) | -2.75 (5.09)

4. Secondary Outcome: Curcumin and Pain
Description: To examine the effects of dietary supplementation with curcumin on pain symptoms (pain scale 0-10 with 10 being the worst)
Time Frame: Baseline and 3 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Curcumin | Placebo
Number analyzed (Participants) | 9 | 8
score on a scale
  Baseline | 0.97 (1.3) | 1.3 (1.7)
  90 Days | 0.2 (0.4) | 1.6 (1.7)

5. Secondary Outcome: Curcumin and Inflammation - Interleukin-6
Description: To examine the effects of dietary supplementation with curcumin on markers of systemic inflammation Interleukin-6 (ng/ml)
Time Frame: From Baseline and 3 months
Measure: Mean (Standard Deviation); unit: (ng/ml)
Arm/Group | Curcumin | Placebo
Number analyzed (Participants) | 9 | 8
(ng/ml)
  Baseline | 3.1 (1.4) | 2.7 (1.7)
  90 Days | 3.4 (1.5) | 3.6 (1.5)

ADVERSE EVENTS:
Time Frame: The adverse events were collected over the whole duration of the study for each participant. In particular, each participant underwent a 12-week study period, during which we monitored for adverse events and noted, if any.
Arm/Group | Curcumin | Placebo
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/8
Other Adverse Events (participants affected / at risk) | 0/9 | 0/8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2016-03-17): https://cdn.clinicaltrials.gov/large-docs/80/NCT03085680/Prot_SAP_000.pdf
  • Informed Consent Form (2019-03-06): https://cdn.clinicaltrials.gov/large-docs/80/NCT03085680/ICF_001.pdf